CLINICAL TRIAL: NCT00033332
Title: A Randomized Phase III Trial Of Thalidomide (NSC # 66847) Plus Dexamethasone Versus Dexamethasone In Newly Diagnosed Multiple Myeloma
Brief Title: Dexamethasone With or Without Thalidomide in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069274; U10CA021115 (NIH); E-E1A00
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2005-11

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Dexamethasone; Pamidronate; Thalidomide; Zoledronic Acid

INTERVENTIONS:
Drug: dexamethasone
Drug: pamidronate disodium
Drug: thalidomide
Drug: zoledronic acid

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. Combining dexamethasone and thalidomide may kill more cancer cells. It is not yet known whether dexamethasone is more effective with or without thalidomide in treating multiple myeloma.

PURPOSE: Randomized phase III trial to determine the effectiveness of dexamethasone with or without thalidomide in treating patients who have multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rate of patients with newly diagnosed multiple myeloma treated with dexamethasone with or without thalidomide.
* Compare the toxicity of these regimens in these patients.
* Assess the effect of thalidomide on bone marrow microvessel density and angiogenesis grade and on the expression of vascular endothelial growth factor and basic fibroblast growth factor in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral thalidomide once daily on days 1-28 and oral dexamethasone once daily on days 1-4, 9-12, and 17-20. Patients also receive either pamidronate IV over 2-4 hours or zoledronate IV over 15 minutes on day 1 for bone strengthening.
* Arm II: Patients receive dexamethasone and pamidronate or zoledronate as in arm I.

Treatment in both arms repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients may receive additional courses after the fourth course at the physician's discretion.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually for 2 years.

PROJECTED ACCRUAL: A total of 194 patients (97 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed symptomatic multiple myeloma confirmed by the following:

  * Bone marrow plasmacytosis with at least 10% plasma cells or sheets of plasma cells or biopsy-proven plasmacytosis
  * Monoclonal protein (M protein) at least 1.0 g/dL on serum protein electrophoresis or at least 200 mg of monoclonal light chain on a 24-hour urine protein electrophoresis
* No smoldering myeloma or monoclonal gammopathy of undetermined significance

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 50,000/mm^3
* Hemoglobin greater than 7 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* ALT and AST no greater than 2.5 times upper limit of normal

Renal:

* Creatinine less than 3 mg/dL

Cardiovascular:

* No prior or concurrent deep venous thrombosis

Other:

* Prior malignancy allowed provided the following criteria are met:

  * Received prior treatment with curative intent
  * Free of disease for the time period appropriate for cure of the specific cancer
* No grade 2 or greater peripheral neuropathy due to other medical conditions
* No active infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 1 highly effective method and 1 additional method of contraception for 1 month before, during, and for 4 weeks after study for women and effective barrier contraception for men during and for 4 weeks after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy for multiple myeloma
* No other concurrent biologic therapy for multiple myeloma

Chemotherapy:

* No prior chemotherapy for multiple myeloma
* No other concurrent chemotherapy for multiple myeloma

Endocrine therapy:

* More than 6 months since prior systemic dexamethasone or glucocorticoids
* No concurrent corticosteroids

Radiotherapy:

* At least 4 weeks since prior palliative, localized radiotherapy
* Concurrent palliative, localized radiotherapy allowed at the physician's discretion

Surgery:

* Not specified

Other:

* No prior systemic therapy for multiple myeloma, except bisphosphonates
* No concurrent anticoagulant therapy for deep vein thrombosis
* No concurrent barbiturates or alcohol (thalidomide arm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-04; Primary Completion 2006-03 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. V. Rajkumar, MD, Study Chair — Mayo Clinic
Locations (78):
- United States (75):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Gainesville, Gainesville, Florida
  - UF Shands Cancer Center, Gainesville, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Tuft-New England Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
- Pretoria Academic Hospitals, Pretoria, South Africa

REFERENCES:
- [Background] Ballester O. The emperor's new clothes or the current practice of clinical trials for multiple myeloma in the USA. Cancer Invest. 2008 Jun;26(5):445-7. doi: 10.1080/07357900701874641. PMID 18568765
- [Background] Johnson DC, Corthals S, Ramos C, Hoering A, Cocks K, Dickens NJ, Haessler J, Goldschmidt H, Child JA, Bell SE, Jackson G, Baris D, Rajkumar SV, Davies FE, Durie BG, Crowley J, Sonneveld P, Van Ness B, Morgan GJ. Genetic associations with thalidomide mediated venous thrombotic events in myeloma identified using targeted genotyping. Blood. 2008 Dec 15;112(13):4924-34. doi: 10.1182/blood-2008-02-140434. Epub 2008 Sep 19. PMID 18805967
- [Result] Kumar S, Greipp PR, Haug JL, et al.: Correlation of bone marrow angiogenesis and response to thalidomide dexamethasone in multiple myeloma. [Abstract] J Clin Oncol 24 (Suppl 18): A-7621, 451s, 2006.
- [Result] Rajkumar SV, Blood E, Vesole D, Fonseca R, Greipp PR; Eastern Cooperative Oncology Group. Phase III clinical trial of thalidomide plus dexamethasone compared with dexamethasone alone in newly diagnosed multiple myeloma: a clinical trial coordinated by the Eastern Cooperative Oncology Group. J Clin Oncol. 2006 Jan 20;24(3):431-6. doi: 10.1200/JCO.2005.03.0221. Epub 2005 Dec 19. PMID 16365178
- [Result] Greipp PR. Eastern Cooperative Oncology Group E1A00: phase III randomized study of dexamethasone with or without thalidomide in patients with newly diagnosed multiple myeloma. Clin Adv Hematol Oncol. 2003 Mar;1(3):188-9. No abstract available. PMID 16224404